CLINICAL TRIAL: NCT06888687
Title: Continuous Glucose Monitoring-Assisted Remote E-health Dietetics to Empower People With Type 2 Diabetes
Brief Title: Comparison of Dietetics Support With and Without Continuous Glucose Monitoring in Individuals With Type 2 Diabetes.
Acronym: CARE-T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian Catholic University (Other)
Collaborators: Abbott Diabetes Care (Industry); University of Adelaide (Other); The University of Queensland (Other); Monash University (Other); University of Melbourne (Other); Deakin University (Other)
Responsible Party: Principal Investigator, Evelyn Parr, Principal Investigator, Australian Catholic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-3690HC
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Continuous Glucose Measurement; Dietary Modification
Keywords: Continual Glucose Monitoring; Type 2 Diabetes; Non-insulin dependant Diabetes; Dietitian Support; Health Behaviours
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietetic support only (Active Comparator): This group is designed to act as a comparator using 'standard care' in dietetics practice. Dietary advice provided to this participant group will be performed by Accredited Practicing Dietitians (APDs) in line with evidence-based guidelines, specifically the T2DM best-practice guidelines plus Australian Dietary Guidelines (i.e. Australian Guide to Healthy Eating) to improve diet quality, and strategies to promote adherence.
  Interventions: Behavioral: Dietetic support
- CGM plus dietetic support (Experimental): The CGM plus dietetic support group will be provided 'standard care' dietetic support alongside the use, and interpretation of, the CGM data collected to assist in the understanding of dietary modifications on glucose management. As per the DIET group, dietary advice provided to this participant group will be performed by Accredited Practicing Dietitians (APDs) in line with evidence-based guidelines, specifically the T2DM best-practice guidelines plus Australian Dietary Guidelines (i.e. Australian Guide to Healthy Eating) to improve diet quality, and strategies to promote adherence. The CGM data collected via LibreLink will be used by both the participant and the dietitian to inform dietary modifications.
  Interventions: Behavioral: Dietetic support; Device: Continuous glucose monitoring

INTERVENTIONS:
Behavioral: Dietetic support — Dietary advice will be provided by Accredited Practicing Dietitians (APDs) in line with evidence-based guidelines, specifically the T2DM best-practice guidelines plus Australian Dietary Guidelines (i.e. Australian Guide to Healthy Eating) to improve diet quality, and strategies to promote adherence.
Device: Continuous glucose monitoring — Abbott FreeStyle Libre 2+ CGM sensors will be used to provide feedback on interstitial glucose concentrations over 15 day periods per sensor.
  Arms: CGM plus dietetic support

SUMMARY:
A parallel, single-blinded, randomised clinical trial conducted remotely across Australia from the Mary MacKillop Institute for Health Research (MMIHR, Australian Catholic University) for individuals with type 2 diabetes, by researchers from Australian Catholic University, University of Adelaide, University of Queensland, University of Wollongong, Monash University, Monash Partners, Deakin University, La Trobe University and Melbourne University.

DETAILED DESCRIPTION:
In a parallel groups design, a total of 156 individuals will be recruited. After baseline pathology (HbA1c), blinded (Libre Pro iQ) continuous glucose monitoring (CGM) data and questionnaires (via REDCap) have been collected, participants will be randomised into one of two groups (DIET, dietetic support only; CGMD, CGM plus dietetic support). All participants will receive four (4) dietetic consults via telehealth at weeks 2, 6, 10 and 16, the content of which will be related to the randomised condition. Measurements will be repeated at 3 and 6 months from baseline to assess the changes in primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years
* Reside anywhere in Australia and have a postal address
* Confirmed T2D diagnosis by a GP/endocrinologist
* Current HbA1c of ≥7.0%
* Have a smartphone and able to independently use it

Exclusion Criteria:

* Under the age of 18 years
* Use of insulin therapy (within the last three months) or medications which interfere with blood glucose levels (i.e. steroids)
* Use of CGM within the last six months
* Eating Disorder Examination Questionnaire (EDE-Q) global score >2.8 OR global score > or equal to 1.52, with sum of Q14-18 > or equal to 4
* Currently having ongoing consultations with an APD or have had a consult with an APD (within last three months)
* Not weight stable (>5 kg change over last three months)
* Severe hypoglycaemic event (i.e. requiring assistance) within last six months
* Change of antihyperglcyaemic medications within last three months
* Women who are pregnant or breastfeeding (within 24 weeks)
* History of psychotic disorder, or current diagnosis of other major psychiatric illness (e.g. mood disorder, eating disorder, substance use disorder)
* History of blood disorders (including but, not limited to, anemia and thalassemia) that impact the primary outcome (HbA1c)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
HbA1c | baseline, 6 months
  Glycated haemoglobin concentration

SECONDARY OUTCOMES:
HbA1c | 3 months
  Glycated haemoglobin concentration
24 h assessment of glycaemia | baseline, 6 months
  24 h glucose measures assessed by blinded CGM (including, but not limited to, time in range, CV)
Fasting blood glucose | baseline, 3 months, 6 months
  fasting blood glucose concentrations
hs-CRP | baseline, 3 months, 6 months
  fasting high sensitive C-Peptide concentrations

OTHER OUTCOMES:
CGM application and use | From 0 to 26 weeks, per 2 week period of sensor use
  number of days of CGM use and interaction with viewing CGM data (via LibreLink); CGMD group ony
Per protocol analysis | 6 months
  Primary analysis of all variables is going to be intention to treat.
  Therefore, secondary analysis will be a per-protocol (PP) analysis. Inclusion in PP analysis will be defined by:
  1. Attendance at ≥3 dietetic consults, within ±10 days of the designated 2-, 6-, 10- and 16-week time points; AND,
  2. Completion of both baseline and 6-month (±10 days) HbA1c blood samples, AND,
  3. Completion of ≥5 days of food records at baseline and 6-months.
Dietary intake | baseline, 3 months, 6 months
  energy and macronutrient composition calculated from food records
Adherence | baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 18 weeks, 20 weeks, 26 weeks
  measures of adherence assessed by self-report (questionnaire)
Fasting cholesterol | baseline, 3 months, 6 months
  Fasting cholesterol concentrations (total, HDL and LDL)
Fasting lipid concentration | baseline, 3 months, 6 months
  fasting triglyceride concentrations
Medication effect score (MES) | baseline, 6 months
  Medication effect score for antihyperglycemic medications
Participant experience | 6 months
  Qualitative semi-structured interviews
Physical activity | baseline, 3 months, 6 months
  Self-reported questionnaire (International Physical Activity Questionnaire (IPAQ) - Long Form)
Sleep quality and quantity | baseline, 3 months, 6 months
  Self-reported questionnaire (Pittsburgh Sleep Quality Index (PSQI))
Eating behaviours | baseline, 3 months, 6 months
  Self-reported questionnaire (Eating Disorders Examination Questionnaire (EDEQ))
Health literacy | baseline, 3 months, 6 months
  self-reported questionnaire (Health Literacy Questionnaire (HLQ))
Dietary quality | baseline, 3 months, 6 months
  Assessed using the Healthy Eating Index For Australian adults (HEIFA)
Diabetes self-management | baseline, 3 months, 6 months
  Self-reported questionnaire (Diabetes Self-Management Questionnaire (DSMQ-R))
Diabetes distress | baseline, 3 months, 6 months
  Self-reported questionnaire (Type 2 Diabetes Distress Assessment Scale (T2DDAS))
Overall well-being | baseline, 3 months, 6 months
  Self-reported questionnaire (WHO-5)
Diabetes-specific well-being | baseline, 3 months, 6 months
  Self-reported questionnaire (DAWN Impact of Diabetes Profile (DIDP-7))
Treatment satisfaction | baseline, 3 months, 6 months
  self-reported questionnaire (Diabetes Treatment Satisfaction Questionnaire (DTSQs (status) and DTSQc (change)))

CONTACTS AND LOCATIONS:
Locations (1):
- Australian Catholic University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding author for a period of 36 months from publication, upon reasonable request for academic use. The data will not be made publicly available, as it contains information that could compromise research participant consent.
Supporting Information: Study Protocol
Access Criteria: Reasonable requests of data for academic use will be considered. Requests can be made to the corresponding author of the publication. Data will not be made publicly available as it contains information that could compromise research participant consent.